CLINICAL TRIAL: NCT02383173
Title: Evaluation of Methods for Implementation of a Comfort Care Order Set
Acronym: BEACON II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 12-071
Record Dates: First submitted 2014-12-23; First posted 2015-03-09 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Terminal Conditions, End of Life
Keywords: end of life; palliative care; implementation
MeSH Terms: conditions — Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic Implementation Approach (Active Comparator): Basic approach to implementing a Comfort Care Education Intervention utilizing the established infrastructure of Palliative Care Consult Teams
  Interventions: Other: Basic Implementation Approach
- Enhanced Implementation Approach (Experimental): Enhanced approach to implementing a Comfort Care Education Intervention utilizing the established infrastructure of Palliative Care Consult Teams
  Interventions: Other: Enhanced Implementation Approach

INTERVENTIONS:
Other: Basic Implementation Approach — Comfort Care Education Intervention utilizing the established infrastructure of Palliative Care Consult Teams, using a Basic Implementation Approach with a teleconference to review educational materials and activate PCCTs to educate other providers.
  Arms: Basic Implementation Approach
Other: Enhanced Implementation Approach — Comfort Care Education Intervention utilizing the established infrastructure of Palliative Care Consult Teams, using an Enhanced Implementation Approach with in-person, train-the-"champion" workshops to prepare PCCT members to be leaders and trainers at their home sites
  Arms: Enhanced Implementation Approach

SUMMARY:
The overarching goal of this research program is to improve the quality of end-of-life care provided to Veterans dying in VA Medical Centers (VAMCs), by transferring the best practices of home hospice and palliative care for the last days and hours of life into the inpatient setting. This trial will examine two methods of delivering a Comfort Care Education Intervention utilizing the established infrastructure of VA Palliative Care Consult Teams (PCCT): a Basic Implementation Approach using a teleconference to review educational materials and activate PCCTs to educate other providers, and an Enhanced Implementation Approach utilizing in-person, train-the-"champion" workshops to prepare PCCT members to be leaders and trainers at their home sites. Findings will provide a robust evaluation of the implementation process, and will be used to refine the Comfort Care Education Intervention and implementation strategies in preparation for nationwide dissemination of best practices for end-of-life care within the VA Healthcare System.

DETAILED DESCRIPTION:
Anticipated Impacts on Veterans' Healthcare: The overarching goal of this research program is to improve the quality of end-of-life care provided to Veterans dying in VA Medical Centers (VAMCs), by transferring the best practices of home hospice and palliative care for the last days and hours of life into the inpatient setting.

Project Background: Often, patients who are near the end of life are not recognized as actively dying. As a result, their suffering may not be appreciated or managed properly, and may even be exacerbated by usual medical care when aggressive, futile, or iatrogenically harmful treatments are continued. During this time, supportive and comfort care treatment plans can be implemented to reduce suffering and improve the quality of care provided to these patients. The investigative team has developed and evaluated an education-based intervention to teach providers how to identify patients who are actively dying and to implement care plans appropriate for the last days or hours of life. To facilitate use of these interventions, an electronic Comfort Care Order Set (CCOS) was designed and integrated into the Computerized Patient Record System (CPRS) to support and guide the selection of comfort care treatments. The effectiveness of the Comfort Care Education Intervention has been demonstrated in 7 VAMCs and it is ready for implementation on a broader scale.

Project Objectives: This trial will extend this line of research by examining two methods of delivering this Comfort Care Education Intervention utilizing the established infrastructure of Palliative Care Consult Teams (PCCT): a Basic Implementation Approach using a teleconference to review educational materials and activate PCCTs to educate other providers, and an Enhanced Implementation Approach utilizing in-person, train-the-"champion" workshops to prepare PCCT members to be leaders and trainers at their home sites. The aims of this study are 1) to compare the effectiveness of the two approaches for changing provider behavior, as reflected in documented processes of end-of-life care, 2) to formatively evaluate PCCT members' experiences with and perceptions of the two approaches, and 3) to quantitatively evaluate PCCT members' perceptions of the training received and its impact on attitudes, skills, and perceived efficacy to care for patients and teach other providers.

Project Methods: PCCTs at 47 VA Medical Centers will be recruited to participate in the trial and randomized to receive the Comfort Care Education Intervention using the Basic or the Enhanced Implementation Approach. Data on processes of end-of-life care will be abstracted from the CPRS medical records of Veterans who die before and after the interventions, including presence of an active opioid order at time of death (primary endpoint), other medication orders and administration, do-not-resuscitate orders, palliative care consult orders, location of death, presence of nasogastric tubes/intravenous lines, restraints, and pastoral care. Semi-structured telephone interviews will be conducted with all participating PCCT members to explore their perceptions of training, the process of teaching other providers at each site, barriers and facilitators they encountered, how prepared they felt to overcome these barriers, and specific needs and preferences regarding the implementation approach.

Findings will provide a robust evaluation of the implementation process, and will be used to refine the Comfort Care Education Intervention and implementation strategies in preparation for nationwide dissemination of best practices for end-of-life care within the VA Healthcare System.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, each provider had to be a member of a VA palliative care consult team (PCCT)

Exclusion Criteria:

VAMCs were excluded if the facility scored in the top 10th percentile or lowest 10th percentile on PROMISE after-death survey; if they had no prescribing provider on the PCCT team; or if there were fewer than 30 deaths in VAMC during the reporting period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Burgio, PhD MA BA, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailey FA, Williams BR, Goode PS, Kennedy RE, Redden DT, Kvale E, Bakitas M, Dionne-Odom JN, Burgio KL. Comparison of Two Methods for Implementing Comfort Care Order Sets in the Inpatient Setting: a Cluster Randomized Trial. J Gen Intern Med. 2021 Jul;36(7):1928-1936. doi: 10.1007/s11606-020-06482-x. Epub 2021 Feb 5. PMID 33547573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Palliative Care Consult Teams (PCCT) from eligible VA Medical Centers were recruited to participate in the education interventions. Demographic characteristics were not collected on providers.
Pre-assignment Details: Eligibility of VAMCs and Palliative Care Consult Team members were determined before enrollment. All those enrolled teams were randomized.
Units Other Than Participants: Palliative Care Consult Teams
Period: Overall Study
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Started | 88; 23 Palliative Care Consult Teams | 46; 24 Palliative Care Consult Teams
Completed | 88; 23 Palliative Care Consult Teams | 44; 23 Palliative Care Consult Teams
Not Completed | 0; 0 Palliative Care Consult Teams | 2; 1 Palliative Care Consult Teams
Not completed — Palliative Care Team withdrew | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants is greater than the number Started in the Participant Flow. The participant flow numbers describe the study participants, VA providers who participated in the education intervention. Data in Baseline Characteristics describe the patients whose medical records were abstracted to measure outcomes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach | Total
Number analyzed (Participants) | 3078 | 3413 | 6491
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 participant is missing age data
  Participants
    number analyzed (Participants) | 3078 | 3412 | 6490
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 645 | 557 | 1202
    >=65 years | 2433 | 2855 | 5288
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant was missing age data
  years
    number analyzed (Participants) | 3078 | 3412 | 6490
    (all) | 74.2 (11.6) | 75.6 (11.4) | 75.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 88 | 165
  Male | 3001 | 3325 | 6326
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 20 | 31
  Asian | 15 | 14 | 29
  Native Hawaiian or Other Pacific Islander | 33 | 16 | 49
  Black or African American | 659 | 751 | 1410
  White | 2096 | 2415 | 4511
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 264 | 197 | 461
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3078 | 3413 | 6491

OUTCOME MEASURES:

1. Primary Outcome: Presence of an Active Opioid Order at Time of Death
Description: presence of an active opioid order at time of death in Veteran's medical record
Time Frame: at time of death for veterans who died in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 1330 | 1543
Statistical Analysis 1: Comparison: Basic Implementation Approach vs Enhanced Implementation Approach; Generalized Estimating Equation (GEE) analyses of post-intervention data were used to account for clustering. We adjusted for age, race, cancer, length of stay and study year; Test type: Other; p = 0.445, Generalized Estimating Equation (GEE); Sandwich estimators were used to adjust for the small number of clusters

2. Secondary Outcome: Presence of an Order for Benzodiazepine Medication
Description: presence of an order for benzodiazepine medication in the last 7 days of life
Time Frame: last 7 days of life for veterans who died in the 9 months following the intervention period
Population: Veterans who died in the 9 months following the intervention period
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 1025 | 1117

3. Secondary Outcome: Presence of a Do-not-resuscitate Order
Description: presence of a do-not-resuscitate order in the last 7 days of life
Time Frame: last 7 days of life for veterans who died in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 1336 | 1504

4. Secondary Outcome: Presence of a Palliative Care Consult Order
Description: presence of a palliative care consult order in the last 7 days of life
Time Frame: last 7 days of life for veterans who died in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 1208 | 1426

5. Secondary Outcome: Location of Death
Description: death in intensive care unit
Time Frame: in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 436 | 408

6. Secondary Outcome: Presence of a Nasogastric Tube
Description: presence of a nasogastric tube at time of death
Time Frame: in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 161 | 141

7. Secondary Outcome: Presence of an Intravenous Line
Description: presence of an intravenous line at time of death
Time Frame: in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 141 | 184

8. Secondary Outcome: Presence of Restraints
Description: presence of restraints at time of death
Time Frame: in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 86 | 73

9. Secondary Outcome: Presence of a Pastoral Care Visit
Description: presence of a pastoral care visit in the last 7 days of life
Time Frame: last 7 days of life for veterans who died in the 9 months following the intervention period
Population: Veterans who died as inpatients in acute care units of VA Medical Centers
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
Number analyzed (Participants) | 1519 | 1687
Participants | 1060 | 1271

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed. All patients were already deceased and outcomes were based on review of their medical records.
Arm/Group | Basic Implementation Approach | Enhanced Implementation Approach
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Analyses limited by baseline values on some key endpoints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02383173/Prot_SAP_000.pdf